CLINICAL TRIAL: NCT02729246
Title: Bariatric Surgery for the Treatment of Type 2 Diabetes - Clinical Effects and Underlying Mechanisms
Acronym: Bariglykos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2014/255
Record Dates: First submitted 2016-03-16; First posted 2016-04-06 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention)
- Surgery Group (Other): The patients in this group will undergo Laparoscopic Gastric Bypass surgery
  Interventions: Procedure: Laparoscopic Gastric Bypass

INTERVENTIONS:
Procedure: Laparoscopic Gastric Bypass
  Arms: Surgery Group

SUMMARY:
The main purpose of this project is to further explore the metabolic effects and the mechanisms underlying the improvement in glucose homeostasis following bariatric surgery. The project will involve both prevention and treatment of Type 2 Diabetes (T2D), and both pre-diabetic as well as diabetic subjects with obesity will be included. This part of the project focuses on patients with manifest T2D and they will be assigned to surgical and non-surgical intervention, respectively, in a strictly controlled and randomized manner.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-60 years
* Type 2 Diabetes Mellitus with duration of no more than 10 years, treated with 0-3 oral anti-diabetic drugs or Glucagon-like peptide-1 (GLP-1) analog.

Exclusion Criteria:

* Pregnant or planning to be pregnant during the study.
* Known or suspected history of significant drug abuse.
* History of alcohol abuse or excessive intake of alcohol as judged by investigator.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator
* Sleep apnea
* Any previous serious cardiovascular event, stroke , acute myocardial infarction.
* Diabetes complications : proliferative retinopathy, maculopathy, chronic renal failure stadium 3 with an Estimated Glomerular Filtration Rate (eGFR) <60, foot ulcers, symptomatic neuropathy
* Medications within 3 months : Insulin, Thiazolidinediones
* Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study and /or for the patients safety
* Judgment by the investigator that the subject should not participate in the study if considers subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10; Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Glucose Turnover | 1 month after surgery
Change from Baseline of homeostatic model assessment (HOMA) for insulin resistance | 1 month after surgery
Change from Baseline of beta cell function | 1 month after surgery

SECONDARY OUTCOMES:
Change from Baseline of Glucose Turnover | 6 months after surgery
Change from Baseline of Glucose Turnover | 24 months after surgery
Change from Baseline of homeostatic model assessment (HOMA) for insulin resistance | 6 months after surgery
Change from Baseline of homeostatic model assessment (HOMA) for insulin resistance | 24 months after surgery
Change from Baseline of beta cell function | 6 months after surgery
Change from Baseline of beta cell function | 24 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eriksson, Professor, Principal Investigator — Department of Medical Sciences, Clinical diabetology and metabolism
Locations (1):
- Uppsala University, Department of Medical Sciences, Clinical diabetology and metabolism, Uppsala, Sweden

REFERENCES:
- [Derived] Almby KE, Katsogiannos P, Pereira MJ, Karlsson FA, Sundbom M, Wiklund U, Kamble PG, Eriksson JW. Time Course of Metabolic, Neuroendocrine, and Adipose Effects During 2 Years of Follow-up After Gastric Bypass in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2021 Sep 27;106(10):e4049-e4061. doi: 10.1210/clinem/dgab398. PMID 34086911
- [Derived] Katsogiannos P, Randell E, Sundbom M, Rosenblad A, Eriksson JW, Leksell J. Quality of life after gastric bypass surgery in patients with type 2 diabetes: patients' experiences during 2 years of follow-up. Diabetol Metab Syndr. 2020 Oct 12;12:90. doi: 10.1186/s13098-020-00597-1. eCollection 2020. PMID 33062061
- [Derived] Katsogiannos P, Kamble PG, Boersma GJ, Karlsson FA, Lundkvist P, Sundbom M, Pereira MJ, Eriksson JW. Early Changes in Adipose Tissue Morphology, Gene Expression, and Metabolism After RYGB in Patients With Obesity and T2D. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2601-2613. doi: 10.1210/jc.2018-02165. PMID 30689903